CLINICAL TRIAL: NCT04969042
Title: Efficacy of Closed-loop Functional Spinal Cord Stimulation on Walking Rehabilitation in Patients With Spinal Cord Injury
Brief Title: Closed-loop Functional Spinal Cord Stimulation in Patients With Spinal Cord Injury
Acronym: COFUN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luming Li (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Sponsor-Investigator, Luming Li, Director of National Engineering Laboratory for Neuromodulation, Tsinghua University
Organization: Tsinghua University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202000325
Record Dates: First submitted 2021-07-06; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Stimulation; Closed-Loop
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stimulation (Experimental): Participants will receive pre-implantation rehabilitation, implantation of the closed-loop spinal cord stimulator, and stimulation (according to the functional mapping) assisted rehabilitation post-implantation during the trial.
  Interventions: Device: Pins Medical G122 RS

INTERVENTIONS:
Device: Pins Medical G122 RS — G122RS model implanted spinal cord stimulation device, which could give closed-loop functional stimulation in the epidural space

SUMMARY:
The purpose of this experiment is to evaluate the efficacy of Closed-loop Functional Spinal Cord Stimulation on Walking Rehabilitation in Patients after Spinal Cord Injury

DETAILED DESCRIPTION:
The whole course will last around 12 months, during which there will be: Pre-implant evaluations and standard rehabilitation (6-10 weeks), Stimulator implantation and stimulation optimization (4-8 weeks), Rehabilitation training with stimulation (6 months). At the end of the protocol, the study aims to make the patients walk better and faster.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~70
* Spinal cord injury staging(AIS) A,B,C or D
* Level of lesion is T10 and above
* Distance between lesion and conus >60mm
* Injured Time > 3 months
* Capable of participating rehabilitation program
* Agree to comply with all conditions of the study and to attend all required study training and visits

Exclusion Criteria:

* With Obvious psychiatric disorder that cannot complete relevant questionaires
* Cognitive impairment
* Severe autonomic reflex disorder
* Severe muscle atrophy and joint contracture
* Cannot participate in spinal cord stimulation surgery or follow-up visits
* Life expectancy less than 12 months
* Abnormal blood or other physiological examinations that cannot conduct surgery, such as blood coagulation disorder or kidney/liver abnormalities
* Uncontrollable hypertension, heart diseases, respiratory diseases or took related medicine in last 3 months
* Unsuitable candidates in PI's perspective

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
WISCI III | Change from Baseline to the 8 month after implantation.
  A Common method used to evaluate SCI patient's walking capability in clinical setting
10-metre Walking Test 10-metre Walking Test 10-metre Walking Test 10 meter wlaking | Change from Baseline to the 8 month after implantation.
  10-Meter Walk Test (10MWT) is commonly used to measure walking speeds during two conditions: a self-selected normal speed, and a self-selected 'faster-than-normal' speed.
Weight Bearing Capacity | Change from Baseline to the 8 month after implantation.
  Weight-bearing capacity (WBC) is an important outcome to monitor and particularly relevant in patients with severe motor impairments who cannot walk independently. The investigators use LPG HUBER360 to examine subjects' weight bearing capacity

CONTACTS AND LOCATIONS:
Overall Officials: Luming Li, PhD, Principal Investigator — National Engineering Laboratory for Neuromodulation
Locations (1):
- National Engineering Laboratory for Neuromodulation, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No